CLINICAL TRIAL: NCT02130700
Title: A Phase 2 Open-Label Study to Evaluate the Efficacy and Safety of VT-464 in Patients With Metastatic Castration Resistant Prostate Cancer Who Have Previously Been Treated With Enzalutamide, Androgen Receptor Positive Triple-Negative Breast Cancer Patients, and Men With ER Positive Breast Cancer
Brief Title: Oral VT-464 in Patients With Castration-Resistant Prostate Cancer Previously Treated With Enzalutamide, Androgen Receptor Positive Triple-Negative Breast Cancer Patients, and Men With ER Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocrin Pharmaceutical (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INO-VT-464-CL-002; VMT-VT-464-CL-002 (Other: Innocrin); NCT02117531 (obsolete NCT alias)
Record Dates: First submitted 2014-04-22; First posted 2014-05-05 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: mCRPC; metastatic; castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — VT-464; seviteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Chemotherapy-Naive Patients (Experimental): VT-464: given orally twice daily in 28-day cycles
  Interventions: Drug: VT-464: given orally twice daily in 28-day cycles
- Previous Chemotherapy Patients (Experimental): VT-464: given orally twice daily in 28-day cycles
  Interventions: Drug: VT-464: given orally twice daily in 28-day cycles
- AR Positive 1 - 9% TNBC (Experimental): VT-464: given orally once daily in 28-day cycles
  Interventions: Drug: VT-464: given orally once daily in 28-day cycles
- Male ER Positive (Experimental): VT-464: given orally once daily in 28-day cycles
  Interventions: Drug: VT-464: given orally once daily in 28-day cycles
- AR Positive >10% TNBC (Experimental): VT-464: given orally once daily in 28-day cycles
  Interventions: Drug: VT-464: given orally once daily in 28-day cycles

INTERVENTIONS:
Drug: VT-464: given orally twice daily in 28-day cycles — Oral VT-464 given twice daily, in continuous 28-day cycles at the recommended Phase 2 dose
  Other Names: VT-464
  Arms: Chemotherapy-Naive Patients; Previous Chemotherapy Patients
Drug: VT-464: given orally once daily in 28-day cycles — Oral VT-464 given once daily, in continuous 28-day cycles at the recommended Phase 2 dose
  Other Names: seviteronel
  Arms: AR Positive 1 - 9% TNBC; AR Positive >10% TNBC; Male ER Positive

SUMMARY:
The goal of this clinical study is to determine the safety and efficacy of VT-464, a lyase-selective inhibitor of CYP17, in patients with castration-resistant prostate cancer (CRPC) who have been previously treated with Enzalutamide, Androgen Receptor Positive Triple-Negative Breast Cancer Patients, and Men with ER positive Breast Cancer.

DETAILED DESCRIPTION:
This is a Phase 2 open-label study of VT-464 in patients with progressive, metastatic castration-resistant prostate cancer (mCRPC) who have been previously treated with enzalutamide, female patients with triple negative, AR positive breast cancer and men with ER positive breast cancer. The study consists of five cohorts: patients in Cohort 1 must have never received prior chemotherapy. Patients in Cohort 2 must have received at least one (and not more) prior course of chemotherapy for CRPC. Women with TNBC will be stratified into two cohorts AR 1 to 9% (cohort 3) and AR > 10% (cohort 4). Cohort 5 will consist of men who have been diagnosed with ER+ breast cancer and have failed at least one prior endocrine therapy.

ELIGIBILITY:
Key Eligibility Criteria:

* Patients must have documented histological or cytological evidence of adenocarcinoma of the prostate.
* Must have progressive, metastatic castration-resistant prostate cancer (mCRPC). There must be radiographic evidence of disease after primary treatment with surgery or radiotherapy that has continued to progress radiographically or biochemically (rising PSA levels on successive measurements) despite adequate androgen-deprivation therapy, which is defined as having undergone bilateral surgical castration or continued treatment on GnRH agonists or antagonists.
* All patients in this trial must have been treated with enzalutamide.
* Patients in Cohort 1 will not be allowed to have received prior chemotherapy; patients in Cohort 2 must have received one (and not more) prior course of chemotherapy for mCRPC.
* Progression must be evidenced and documented by any of the following parameters:

  * PSA progression defined by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination
  * Appearance of one or more new lesions on bone scan
  * Progressive measurable disease by RECIST 1.1

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The change in PSA from baseline using waterfall plots in response to 12-weeks of treatment with VT-464 | 12 weeks
  To determine the PSA response as defined by a ≥ 50% decrease in serum PSA per the Prostate Cancer Clinical Trials Working Group 2 criteria after each cycle and after 12 weeks of dosing with VT-464 compared to PSA level at baseline in patients who have been previously treated with enzalutamide.
Progression-free survival using Kaplan-Meier curves | 8 months
  Kaplan-Meier curves of progression-free survival (PFS) will be constructed in each cohort and the median PFS will be determined and informally compared to any available results.
Determine clinical benefit rate (CBR) as defined by complete response (CR), partial response (PR) or stable disease (SD) in women with androgen receptor (AR) positive, triple-negative breast cancer | 16 weeks
  Clinical benefit rate will be measured at designated timepoints as listed per protocol
Determine clinical benefit rate (CBR) as defined by complete response (CR), partial response (PR) or stable disease (SD) in women with androgen receptor (AR) positive, triple-negative breast cancer | 24 weeks
  Clinical benefit rate will be measured at designated timepoints as listed per protocol

SECONDARY OUTCOMES:
Overall survival using Kaplan-Meier curves | 32 months
  Overall Survival: will be analyzed similarly to PFS, with a separate Kaplan-Meier curve for each arm. A patient for whom there is no death event will be censored; the censored date will be the date of last contact.
The safety and tolerability of VT-464 by evaluating adverse events, vital signs, physical examination findings, concomitant medications and laboratory tests. | 8 months
  The safety of VT-464 will be evaluated by laboratory evaluation, electrocardiogram, the report of adverse events and concomitant medications at each 28-day cycle of treatment and 4-5 weeks after therapy has been discontinued.
Maximum PSA response compared to baseline | 8 months
  Maximum PSA response will be descriptive in nature and presented for each cohort as a percent of patients and as a waterfall plot.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health, National Cancer Institute, Bethesda, Maryland, United States